CLINICAL TRIAL: NCT02780505
Title: Assessment of the Effect of Vitamin C on Anemia in Patients With Continuous Ambulatory Peritoneal Dialysi
Brief Title: Assessment of the Effect of Vitamin C on Anemia in Patients With Continuous Ambulatory Peritoneal Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad mahdi Sagheb, associate professor of internal medicine ,Nephrology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT905933
Record Dates: First submitted 2016-05-18; First posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin c (Active Comparator): vitamin C supplement orally up to 250 mg per day for 6 weeks was prescribed. Plasma levels of vitamin C and other clinical parameters including hemoglobin, ferritin, TIBC, iron and CRP were measured at the beginning and end of the study.
  Interventions: Drug: vitamin c
- placebo (Placebo Comparator): ُPlacebo prescribed to Group B. Plasma levels of vitamin C and other clinical parameters including hemoglobin, ferritin, TIBC, iron and CRP were measured at the beginning and end of the study
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vitamin c — In the current prospective, double-blind, and randomized trial, 66 patients with peritoneal dialysis were enrolled, and 43 patients were detected with serum vitamin C level below 4 μg/ml to determine the effect of vit C on anemia in patients on CAPD.
  The measured clinical parameters including plasma vitamin C level, hemoglobin (Hb), Ferritin, total iron-binding capacity (TIBC), serum Fe, C-reactive protein (CRP), and transferrin saturation. Consumption of vitamin supplements such as vitamin C (or any other form of it) either oral or parenteral were discontinued three weeks before collecting the samples.
  Other Names: ascorbic acid
  Arms: vitamin c
Drug: placebo — Active (ascorbic acid 250 mg) and placebo (same weight of starch) tablets were similar in shape and size for both study and control groups. Intravenous intervention was not advantageous for hemodialysis subjects and it was impossible for PD patients, therefore, oral administration was used. All follow-up records were stored.
  The erythropoietin (EPO) injections was prescribed for each patient in weekly dose, started one month before collecting blood samples for vitamin C measurement.
  Arms: placebo

SUMMARY:
Among patients with chronic kidney disease (CKD), there is association between anemia and increased chance of mortality mainly because of cardiovascular diseases and stroke, risk of hospitalization, and death prevalence in predialysis patients. Vitamin C plays an important role in iron metabolism and application for red blood cell formation. Infusion of ascorbate supplementation can reduce oxidative stress among hemodialysis patients. This study aimed to assess the effect of vitamin C on patients with continuous ambulatory peritoneal dialysis (CAPD).

DETAILED DESCRIPTION:
World Health Organization (WHO) defines anemia as hemoglobin (Hgb) concentration less than 12.0 g/dL in pre-menopausal women, and lower than 13.0 g/dL in adult males and post-menopausal women .Diagnosis of anemia is of high significance, as it might be the first manifestation of a serious illness. Some chronic diseases which also can lead to anemia: autoimmune disorders, liver cirrhosis, cancer, and chronic renal disease Anemia is associated with poor prognosis of patients with chronic renal disease, especially those undergoing long-term hemodialysis. In patients with Glomerular filtration rate (GFR) less than 25 to 30 mL/min , anemia is observed within 90 percent of patients .

Among patients with chronic kidney disease (CKD), there is association between anemia and increased mortality secondary to cardiovascular diseases Ascorbic acid level is conflicted in under dialysis patients with different ranges of low, normal, and even above normal. In most hemodialysis patients, administration of 150 to 200 mg of vitamin C per day is recommended to maintain its levels. Ascorbic acid or vitamin C increases the delivery of iron from ferritin and the reticuloendothelial system and therefore elevates iron use during heme synthesis.

Vitamin deficiency is one of the cause of increased mortality among hemodialysis patients. During the dialysis process, vitamins are eliminated through hemodialyzer membranes, thus affect red blood cell production .Vitamin C deficiency may play an important role in increased inflammatory status of the dialysis patients . This vitamin has anti-inflammatory effects due to its electron transfer ability.

Several studies have shown the role of vitamins such as vitamin D and B12 in treatment of anemia in patients undergoing hemodialysis .The infusion of ascorbate supplementation might reduce oxidative stress. In addition, vitamin C plays an important role in iron metabolism and application in red blood cell formation . Permeable membrane is highly associated with a significant loss of vitamin C, and this vitamin improve oxidative stress in hemodialysis patients .

We aimed to assess the effect of vitamin C on patients with continuous ambulatory peritoneal dialysis (CAPD).

ELIGIBILITY:
Inclusion Criteria:

1. Long-term treatment of PD (at least more than three months)
2. Hemoglobin less than 15 milligrams per liter
3. Age over 18 years
4. vitamin c level less than 4microgram\ml

Exclusion Criteria:

1. Acute illness (including infectious diseases and cancer) within 3 months prior to determining the level of vitamin C
2. Any recent blood transfusion, recurrent bleeding or hemolysis
3. Supplementation with vitamin C) during the 3 weeks prior to the determination of serum levels 4 -Consumption of tetracycline, antacid and Cholestyramine

5- diagnosis of primary hyperoxaloria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
level of vitamin c hemoglobin | six weeks prescription

SECONDARY OUTCOMES:
c reactive protein | six weeks after prescription

CONTACTS AND LOCATIONS:
Overall Officials: zahra lotfi, fellowship, Principal Investigator — Shiraz University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided